CLINICAL TRIAL: NCT06276257
Title: Comparison Between Paravertebral Block and Usual Analgesia in Patients Undergoing Unilateral Total Mastectomy with Immediate Reconstruction
Brief Title: Paravertebral Block for Mastectomy with Immediate Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-7301
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paravertebral block (Experimental): Preoperative paravertebral block on the side of mastectomy in addition to usual analgesia.
  Interventions: Procedure: Paravertebral block
- Usual analgesia (Active Comparator): Usual analgesia, as per anesthesiologist's preferences.
  Interventions: Procedure: Usual analgesia

INTERVENTIONS:
Procedure: Paravertebral block — An ultrasound-guided technique will be used to inject a volume of 40 mL of ropivacaine 0.2%, up to a maximum of 1.5 mg/kg, into the paravertebral space between the T3 and T4 vertebrae.
  Arms: Paravertebral block
Procedure: Usual analgesia — The patient will receive analgesia as per the anesthesiologist's preferences.
  Arms: Usual analgesia

SUMMARY:
Following a mastectomy, patients may develop chronic pain, called post-mastectomy pain syndrome (PMPS). This syndrome manifests itself as complex neuropathic pain that seems linked to nerve damage suffered either during surgery, during healing or by nervous system dysfunction. However, the exact pathophysiology remains unknown. Typically, the pain is located on the ipsilateral side of the surgery and projects to the anterior thorax to the lateral thorax and may affect the proximal part of the arm. This pain persists for more than three months following the procedure and has the characteristics of neuropathic pain: burning sensation, tingling, electric shock, hyperalgesia, etc. The prevalence of PMDS varies between 2% and 78%; this disparity comes from the fact that there are no clear criteria in the literature for making the diagnosis. One of the risk factors for developing PMDS is the presence of acute pain immediately postoperatively.

The main objective of this study is to compare two analgesic modalities, namely BPV (study modality) and usual analgesia (control modality), in patients undergoing total mastectomy with immediate reconstruction under general anesthesia with the aim of to evaluate their functional pain score at 24, 48 and 72 hours following the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* woman scheduled for unilateral mastectomy with immediate reconstruction

Exclusion Criteria:

* Patients who will have an axillary dissection during surgery.
* Woman with severe hepatic insufficiency (Child Pugh Classification B and above24).
* Woman with kidney failure stage 4 and above25.
* Body mass index (BMI) > 40 kg/m2.
* Woman with an allergy to local anesthetics.
* Woman with a bleeding disorder in whom BPV is contraindicated.
* Woman in whom stopping antiplatelet or anticoagulant therapy does not allow compliance with the standards of practice of neuraxial anesthesia issued by the American Society of Regional Anesthesia.
* Woman with a single lung.
* Pregnant woman.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative pain using the BPI | 24 hours, 28 hours, 72 hours after surgery
  Postoperative pain will be measured using the Brief Pain Inventory (BPI)

SECONDARY OUTCOMES:
Total use of opioids received intraoperatively. | within 3 months after surgery
  Total dose of narcotics received intraoperatively (in mg morphine equivalent)
Use of non-opioid analgesia intraoperatively | During surgery
  Analgesics other than opioids used intraoperatively
Total dose of opioids received in the PACU | During PACU stay
  Total dose of narcotics received in the post-anesthesia care unit (PACU) (in mg morphine equivalent)
Time before first opioid | Within 3 months after surgery
  Time to first opioid dose after surgery
Total opioids consumed in the 48 hours following surgery | Within 48 hours after surgery
  Total quantity of opioids consumed in the 48 hours following surgery (in morphine equivalent)
Chronic pain | At 3 months after surgery
  Presence of chronic pain at the surgical site at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Quebec - Universite Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided